CLINICAL TRIAL: NCT00607919
Title: A Double-Blind Placebo Controlled Study of Atomoxetine Hydrochloride for the Treatment of ADHD in Children and Adolescents With ADHD and Comorbid Dyslexia
Brief Title: Treatment of ADHD With Atomoxetine in Children & Adolescents With ADHD & Comorbid Dyslexia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11672; B4Z-US-LYEB (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Results first posted 2011-12-15 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-11

CONDITIONS: Attention Deficit Hyperactivity Disorder; Dyslexia
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Dyslexia | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atomoxetine (Experimental): Atomoxetine will be administered at 1.0 to 1.4 milligram/kilogram/day (mg/kg/day) given orally once daily in the morning. All eligible patients who complete the double-blind study period will have the option of participating in a 16-week open-label extension period in which patients will be treated with atomoxetine
  Interventions: Drug: Atomoxetine
- Placebo (Placebo Comparator): Placebo will be packaged in the same way as experimental drug to enforce double-blind study design. Placebo will be administered orally once daily in the morning. All eligible patients who complete the double-blind study period will have the option of participating in a 16-week open-label extension period in which patients will be treated with atomoxetine.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine — Atomoxetine will be administered at 1.0 to 1.4 mg/kg/day given orally once daily in the morning for 16 to 32 weeks
  Other Names: LY139603
  Arms: Atomoxetine
Drug: Placebo — oral, daily, for 16 weeks
  Arms: Placebo

SUMMARY:
This study will evaluate the effect of atomoxetine in treating Attention-Deficit/Hyperactivity Disorder (ADHD) symptoms in children and adolescents with ADHD and comorbid reading disability (dyslexia)

ELIGIBILITY:
Inclusion Criteria:

* patients must meet Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) criteria for Attention-Deficit/Hyperactivity Disorder (ADHD)
* patients must achieve a score of 80 or more on the Full Scale Intelligence Quotient
* child or adolescent patients must be 10 to 16 years old
* must be able to communicate in English
* must be able to swallow capsules
* be reliable to keep appointments for clinic visits and all related tests

Exclusion Criteria:

* patients who weigh less than 25 Kg or greater than 70 Kg
* patients with a history of alcohol or drug abuse on a repeated basis within the past 3 months
* patients with documented history of autism, Asperger's syndrome or pervasive developmental disorder
* females who are pregnant or breastfeeding
* patients with a history of severe allergy to more than one class of medications
* patients with documented history of bipolar I or bipolar II disorder, or psychosis

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 209 (Actual)
Dates: Start 2008-03; Primary Completion 2010-11 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (16):
- United States (16):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Irvine, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palo Alto, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Francisco, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Haven, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Libertyville, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chapel Hill, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbus, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burlington, Vermont
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Spokane, Washington

REFERENCES:
- [Derived] McBurnett K, Clemow D, Williams D, Villodas M, Wietecha L, Barkley R. Atomoxetine-Related Change in Sluggish Cognitive Tempo Is Partially Independent of Change in Attention-Deficit/Hyperactivity Disorder Inattentive Symptoms. J Child Adolesc Psychopharmacol. 2017 Feb;27(1):38-42. doi: 10.1089/cap.2016.0115. Epub 2016 Nov 15. PMID 27845858
- [Derived] Shaywitz S, Shaywitz B, Wietecha L, Wigal S, McBurnett K, Williams D, Kronenberger WG, Hooper SR. Effect of Atomoxetine Treatment on Reading and Phonological Skills in Children with Dyslexia or Attention-Deficit/Hyperactivity Disorder and Comorbid Dyslexia in a Randomized, Placebo-Controlled Trial. J Child Adolesc Psychopharmacol. 2017 Feb;27(1):19-28. doi: 10.1089/cap.2015.0189. Epub 2016 Jul 13. PMID 27410907
- [Derived] Bangs ME, Wietecha LA, Wang S, Buchanan AS, Kelsey DK. Meta-analysis of suicide-related behavior or ideation in child, adolescent, and adult patients treated with atomoxetine. J Child Adolesc Psychopharmacol. 2014 Oct;24(8):426-34. doi: 10.1089/cap.2014.0005. Epub 2014 Jul 14. PMID 25019647
- [Derived] Wietecha L, Williams D, Shaywitz S, Shaywitz B, Hooper SR, Wigal SB, Dunn D, McBurnett K. Atomoxetine improved attention in children and adolescents with attention-deficit/hyperactivity disorder and dyslexia in a 16 week, acute, randomized, double-blind trial. J Child Adolesc Psychopharmacol. 2013 Nov;23(9):605-13. doi: 10.1089/cap.2013.0054. Epub 2013 Nov 9. PMID 24206099
- See also: (Lilly Clinical Trial Registry) — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study comprised a 16-week placebo-controlled, double-blind acute phase and followed by an optional 16-week open-label in which all participants were treated with Atomoxetine.
Groups:
- Atomoxetine/Atomoxetine: Participants were assigned to Atomoxetine treatment in both acute and open-label phase
  Atomoxetine was administered at 1.0 to 1.4 milligram/kilogram/day (mg/kg/day) given orally once daily in the morning for 16 weeks. All eligible participants who completed the double-blind acute phase had the option of participating in a 16-week open-label extension period in which participants were treated with Atomoxetine
- Placebo/Atomoxetine: Participants were assigned to placebo in acute phase and Atomoxetine in open-label phase.
  Placebo was packaged in the same way as Atomoxetine, and administered orally once daily in the morning for 16 weeks. All eligible participants who completed the double-blind acute phase had the option of participating in a 16-week open-label extension period in which participants were treated with Atomoxetine
Period: Acute Phase
Arm/Group | Atomoxetine/Atomoxetine | Placebo/Atomoxetine
Started | 120 | 89
Completed | 86 (2 participants completed acute phase but did not continue into open-label.) | 73 (2 participants completed acute phase but did not continue into open-label.)
Not Completed | 34 | 16
Not completed — Adverse Event | 9 | 2
Not completed — Entry Criteria Not Met | 1 | 1
Not completed — Lack of Efficacy | 1 | 2
Not completed — Lost to Follow-up | 9 | 3
Not completed — Parent/Caregiver Decision | 6 | 4
Not completed — Protocol Violation | 5 | 1
Not completed — Withdrawal by Subject | 3 | 3
Period: Open-Label Phase
Arm/Group | Atomoxetine/Atomoxetine | Placebo/Atomoxetine
Started | 84 | 71
Completed | 74 | 59
Not Completed | 10 | 12
Not completed — Adverse Event | 1 | 5
Not completed — Lost to Follow-up | 4 | 1
Not completed — Protocol Violation | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Parent/Caregiver Decision | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Atomoxetine/Atomoxetine: Participants were assigned to Atomoxetine treatment in both acute and open-label phase
  Atomoxetine was administered at 1.0 to 1.4 mg/kg/day given orally once daily in the morning for 16 weeks. All eligible participants who completed the double-blind acute phase had the option of participating in a 16-week open-label extension period in which participants were treated with Atomoxetine
- Total: Total of all reporting groups
Arm/Group | Atomoxetine/Atomoxetine | Placebo/Atomoxetine | Total
Number analyzed (Participants) | 120 | 89 | 209
Age Continuous [Mean (Standard Deviation); unit: years] | 12.24 (1.72) | 12.44 (1.90) | 12.32 (1.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 34 | 80
  Male | 74 | 55 | 129
Race/Ethnicity, Customized [Number; unit: participants]
  African | 13 | 11 | 24
  Caucasian | 86 | 66 | 152
  East Asian | 2 | 1 | 3
  Hispanic | 18 | 11 | 29
  West Asian | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 120 | 89 | 209

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Attention-Deficit/Hyperactivity Disorder Rating Scale (ADHDRS) Total Score - Parent Version at Week 16 Endpoint
Description: Measures the 18 symptoms contained in the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR) diagnosis of Attention-Deficit/Hyperactivity Disorder (ADHD). Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often). Total scores range from 0-54. Least Square mean of change from baseline in ADHDRS is from a restricted maximum likelihood-based, mixed model repeated measures analysis which includes the effects of treatment, investigative site, baseline, visit, treatment-by-visit interaction, and baseline-by-visit interaction.
Time Frame: Baseline, 16 weeks
Population: All randomized participants with a baseline and at least one post-baseline result.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- ADHD+ Dyslexia (D): Atomoxetine: Participants with attention-deficit/hyperactivity disorder and comorbid dyslexia (ADHD+D) treated with Atomoxetine
  Atomoxetine was administered at 1.0 to 1.4 mg/kg/day given orally once daily in the morning for 16 weeks. All eligible participants who completed the double-blind acute phase had the option of participating in a 16-week open-label extension period in which participants were treated with Atomoxetine
- ADHD+ Dyslexia (D): Placebo: Participants with attention-deficit/hyperactivity disorder and comorbid dyslexia (ADHD+D) treated with Placebo
  Placebo was packaged in the same way as Atomoxetine, and administered orally once daily in the morning for 16 weeks. All eligible participants who completed the double-blind acute phase had the option of participating in a 16-week open-label extension period in which participants were treated with Atomoxetine
Arm/Group | ADHD+ Dyslexia (D): Atomoxetine | ADHD+ Dyslexia (D): Placebo
Number analyzed (Participants) | 47 | 54
units on a scale | -20.01 (1.45) | -12.27 (1.41)
Statistical Analysis 1: Comparison: ADHD+ Dyslexia (D): Atomoxetine vs ADHD+ Dyslexia (D): Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

2. Secondary Outcome: Change From Baseline in Attention-Deficit/Hyperactivity Disorder Rating Scale (ADHDRS) Total and Subscores - Parent Version at Week 16 Endpoint
Description: The ADHDRS-IV-Parent is an 18-item scale with 1 item for each of the 18 symptoms contained in the DSM-IV diagnosis of ADHD. Each item is scored on a 0 to 3 scale: 0=none (never or rarely); 1=mild (sometimes); 2=moderate (often); 3=severe (very often). Hyperactivity-impulsivity scores range 0-27, and inattention scores range 0-27. Total scores range from 0-54. Higher scores indicate higher impairment.
Time Frame: Baseline, 16 weeks
Population: All randomized participants with a baseline and at least one post-baseline result, and last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- ADHD Alone: Atomoxetine: Participants with attention-deficit/hyperactivity disorder (ADHD) alone treated with Atomoxetine.
  Atomoxetine was administered at 1.0 to 1.4 mg/kg/day given orally once daily in the morning for 16 weeks. All eligible participants who completed the double-blind acute phase had the option of participating in a 16-week open-label extension period in which participants were treated with Atomoxetine
Arm/Group | ADHD+ Dyslexia (D): Atomoxetine | ADHD+ Dyslexia (D): Placebo | ADHD Alone: Atomoxetine
Number analyzed (Participants) | 62 | 58 | 27
units on a scale
  Hyperactivity-Impulsivity Score | -8.23 (5.90) | -5.18 (6.01) | -6.26 (5.10)
  Inattention Score | -10.64 (7.59) | -7.79 (6.52) | -10.33 (7.95)
  Total Score | -18.87 (11.68) | -12.98 (10.75) | -16.59 (11.31)

3. Secondary Outcome: Change From Baseline in Attention-Deficit/Hyperactivity Disorder Rating Scale (ADHDRS) Total and Subscores - Teacher Version at Week 16 Endpoint
Description: The ADHDRS-IV-Teacher is an 18-item scale with 1 item for each of the 18 symptoms contained in the DSM-IV diagnosis of ADHD. Each item is scored on a 0 to 3 scale: 0=none (never or rarely); 1=mild (sometimes); 2=moderate (often); 3=severe (very often). Hyperactivity-impulsivity scores range from 0-27, and inattention scores range from 0-27. Total scores range from 0-54. Higher scores indicate higher impairment.
Time Frame: Baseline, 16 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADHD+ Dyslexia (D): Atomoxetine | ADHD+ Dyslexia (D): Placebo | ADHD Alone: Atomoxetine
Number analyzed (Participants) | 21 | 22 | 11
units on a scale
  Hyperactivity-Impulsivity Score | -2.71 (3.98) | -1.99 (6.54) | -0.82 (4.92)
  Inattention Score | -4.48 (5.17) | -0.99 (5.33) | -2.27 (5.24)
  Total Score | -7.19 (6.83) | -2.98 (10.83) | -3.09 (9.21)

4. Secondary Outcome: Change From Baseline in Woodcock-Johnson III Scores at Week 16 Endpoint
Description: The Woodcock Johnson Tests of Achievement has a Standard Battery (Tests 1-12) of a broad set of scores and an Extended Battery (Tests 13-22) on specific academic strengths and weaknesses. Tests associated with reading skills (1, 2, 7, 9, 13, 17, 20) were administered. Scores for each individual test can range from 0 to over 200 where anything 69 and below is very low and anything 131 and above is very superior. Higher scores indicate better reading skills.
Time Frame: Baseline, 16 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADHD+ Dyslexia (D): Atomoxetine | ADHD+ Dyslexia (D): Placebo | ADHD Alone: Atomoxetine
Number analyzed (Participants) | 51 | 55 | 22
units on a scale
  Basic Reading Skills (Tests 1, 13) | 1.75 (6.04) | 0.87 (6.75) | -0.41 (7.99)
  Letter-Word Identification (Test 1) | 1.18 (7.20) | -0.07 (6.63) | -0.32 (8.04)
  Passage Comprehension (Test 9) | -0.92 (11.43) | -1.02 (8.94) | -4.50 (9.04)
  Reading Comprehension (Test 9, 17) | -0.08 (9.68) | -1.09 (8.81) | -5.00 (7.45)
  Reading Fluency (Test 2) | -0.24 (7.91) | -0.11 (9.19) | 1.36 (8.77)
  Reading Vocabulary (Test 17) | 0.51 (8.92) | -0.16 (9.45) | -3.95 (8.60)
  Spelling (Test 7) | -0.22 (7.32) | -4.16 (12.13) | -0.41 (5.68)
  Spelling of Sounds (Test 20) | 5.67 (16.07) | 3.31 (13.49) | 8.45 (19.78)
  Word Attack (Test 13) | 2.27 (6.75) | 1.13 (9.75) | -0.36 (7.88)

5. Secondary Outcome: Change From Baseline in Comprehensive Test of Phonological Processing (CTOPP) at Week 16 Endpoint
Description: The CTOPP assesses phonological awareness, phonological memory, and rapid naming and is appropriate for ages 7 to 24. The test contains six core subtests. The composite scores are 1) Phonological Awareness, comprised of the standard scores of the Elision and Blending Words; 2) Phonological Memory, comprised of standard scores for Memory for Digits and Non-word Repetition; and 3) Rapid Naming, comprised of standard scores for Rapid Digit Naming and Rapid Letter Naming. Standard scores range from 1-20, and composite scores range from 35-165. Higher scores are better.
Time Frame: Baseline, 16 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADHD+ Dyslexia (D): Atomoxetine | ADHD+ Dyslexia (D): Placebo | ADHD Alone: Atomoxetine
Number analyzed (Participants) | 51 | 55 | 22
units on a scale
  Blending Words | 0.96 (1.90) | 0.95 (1.97) | 1.86 (1.86)
  Elision | 0.88 (2.18) | -0.24 (2.34) | 0.27 (1.91)
  Memory for Digits | 0.47 (2.16) | 0.13 (1.76) | -0.50 (1.90)
  Non-word Repetition | 0.57 (1.79) | 0.51 (2.00) | 0.82 (2.52)
  Phonological Awareness | 5.20 (9.49) | 2.00 (9.34) | 6.82 (11.50)
  Phonological Memory | 2.22 (10.61) | 0.96 (10.16) | 1.36 (11.33)
  Rapid Digit Naming | 0.26 (2.06) | 0.16 (1.75) | 0.23 (1.23)
  Rapid Letter Naming | 0.31 (1.76) | 0.24 (1.64) | 0.14 (1.52)
  Rapid Naming | 1.06 (11.00) | 0.35 (9.75) | -0.59 (10.83)

6. Secondary Outcome: Change From Baseline in Gray Oral Reading Test-4 (GORT-4) at Week 16 Endpoint
Description: The GORT-4 is a norm-referenced test of oral reading rate, accuracy, fluency, and comprehension valid for individuals aged 6 to 18 years old. The test has two parallel forms, Form A and Form B, that are administered in an alternating fashion (e.g. Week 0-Form A, Week 16-Form B, Week 32-Form A.) with each containing 14 separate stories and 5 multiple-choice comprehension questions for each story. GORT-4 yields the following scores: rate, accuracy, fluency, comprehension, and overall reading ability. Standard scores range from 1-20. Higher scores indicate better reading skills.
Time Frame: Baseline, 16 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADHD+ Dyslexia (D): Atomoxetine | ADHD+ Dyslexia (D): Placebo | ADHD Alone: Atomoxetine
Number analyzed (Participants) | 51 | 55 | 21
units on a scale
  Accuracy Score | 0.71 (2.22) | 0.40 (2.02) | 0.95 (2.16)
  Comprehension Score | 0.37 (2.35) | 0.65 (2.50) | -0.33 (1.93)
  Fluency Score | 0.78 (2.81) | 0.33 (2.82) | 1.14 (2.94)
  Oral Reading Quotient | -1.43 (23.34) | 2.87 (20.43) | 2.43 (10.93)
  Rate Score | 0.20 (1.65) | 0.05 (1.54) | 0.38 (2.27)

7. Secondary Outcome: Change From Baseline in Test of Word Reading Efficiency (TOWRE) at Week 16 Endpoint
Description: The TOWRE is a measure of an individual's ability to pronounce printed words accurately and fluently and is appropriate for individuals aged 6 to 24 years old. The TOWRE contains two subtests: Sight Word Efficiency (SWE) which assesses the number of real printed words that can be accurately identified within 45 seconds and Phonemic Decoding Efficiency (PDE) which measures the number of pronounceable printed non-words that can be accurately decoded within 45 seconds. Scores range from 45-146. Higher scores indicate higher reading proficiency.
Time Frame: Baseline, 16 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADHD+ Dyslexia (D): Atomoxetine | ADHD+ Dyslexia (D): Placebo | ADHD Alone: Atomoxetine
Number analyzed (Participants) | 61 | 57 | 26
units on a scale
  Phonemic Decoding Efficiency | 1.92 (6.01) | 1.21 (5.19) | 1.77 (6.78)
  Sight Word Efficiency | 1.38 (5.78) | 1.19 (4.80) | 0.69 (8.84)
  Total Word Reading Efficiency Standard Score | -0.57 (21.98) | 2.81 (11.90) | -5.88 (25.98)

8. Secondary Outcome: Change From Baseline in Working Memory Test Battery for Children (WMTB-C) at Week 16 Endpoint
Description: WMTB-C is assessment of working memory capacities, consisting of 9 subtests (Trials Correct Scores [Range from 55-145], Higher scores are better) reflecting 3 main components of working memory: central executive (CE) control/regulation of working memory (Backward Digit Recall, Listening Recall, Counting Recall); phonological loop (PL) responsible for holding verbal information for short periods (Digit Recall, Word List Matching, Word List Recall, Non-word List Recall); and visuo-spatial sketchpad (VSSP) which holds information in visual and spatial form (Block Recall, Mazes Memory).
Time Frame: Baseline, 16 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADHD+ Dyslexia (D): Atomoxetine | ADHD+ Dyslexia (D): Placebo | ADHD Alone: Atomoxetine
Number analyzed (Participants) | 54 | 56 | 23
units on a scale
  Phonological Loop Component Score (n=51, 54, 21) | 3.57 (10.79) | 1.63 (9.00) | 2.24 (9.78)
  Central Executive Component Score (n=41, 44,12) | 7.34 (10.65) | -0.89 (13.65) | 2.17 (11.77)
  Visuo-Spatial Sketchpad Score (n=47, 43, 21) | 4.15 (11.96) | -0.47 (12.85) | 3.67 (10.77)
  Digit Recall (n=54, 56, 23) | 0.17 (3.42) | 0.55 (3.01) | 0.22 (4.45)
  Word List Matching (n=54, 56, 23) | -0.20 (7.08) | 0.05 (8.65) | 2.04 (9.24)
  Word List Recall (n=54, 56, 23) | 1.00 (3.29) | 0.02 (3.15) | 0.35 (2.98)
  Non-Word List Recall (n=53, 56, 23) | 0.89 (2.74) | 0.71 (2.20) | 0.43 (3.53)
  Block Recall (n=54, 56, 23) | -0.37 (4.20) | -0.80 (4.18) | 0.70 (4.24)
  Mazes Memory (n=54, 56, 23) | 1.94 (5.90) | 1.18 (5.94) | 0.78 (7.33)
  Listening Recall (n=54, 56, 23) | 1.52 (3.32) | 1.00 (3.77) | 0.04 (5.90)
  Counting Recall (n=54, 56, 23) | 0.50 (4.63) | 0.45 (5.07) | 0.48 (5.41)
  Backward Digit Recall (n=54, 56, 23) | 1.30 (3.87) | 0.16 (3.62) | 1.26 (4.20)

9. Secondary Outcome: Change From Baseline in Life Participation Scale-child (LPS-C) Score at Week 16 Endpoint
Description: LPS-C is a short (24 item, 0-3 points per item) parent-rated scale that is designed to assess changes in adaptive functioning related to treatment for ADHD. This scale measures improvements in social, emotional, cognitive, educational, and affiliative (family, friends) functioning, which indirectly reflect improvements in executive functioning. Happy/social subscores range from 0-18, and self-control subscores range from 0-54. Total scores range from 0-72. Higher scores are better for LPS.
Time Frame: Baseline, 16 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADHD+ Dyslexia (D): Atomoxetine | ADHD+ Dyslexia (D): Placebo | ADHD Alone: Atomoxetine
Number analyzed (Participants) | 58 | 57 | 26
units on a scale
  LPS Happy/Social Score | 0.57 (4.19) | 0.53 (4.80) | 1.38 (3.73)
  LPS Self Control Score | 6.06 (8.54) | 4.29 (10.60) | 7.49 (8.46)
  LPS Total Score | 6.51 (11.61) | 4.82 (14.20) | 9.05 (10.63)

10. Secondary Outcome: Change From Baseline in Kiddie Sluggish Cognitive Tempo (K-SCT) at Week 16 Endpoint
Description: The K-SCT rating scale contains 3 components: Youth, Parent, and Teacher ratings. It queries 17 candidate SCT symptoms, such as daydreams, lost in a fog, sluggish/drowsy. Scores range from 0-51. Lower scores indicate less sluggish.
Time Frame: Baseline, 16 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADHD+ Dyslexia (D): Atomoxetine | ADHD+ Dyslexia (D): Placebo | ADHD Alone: Atomoxetine
Number analyzed (Participants) | 56 | 57 | 23
units on a scale
  Total Score-Parent Variation (n= 56, 57, 23) | -7.82 (10.98) | -4.64 (9.67) | -8.24 (9.90)
  Total Score-Teacher Variation (n= 22, 22, 11) | -8.82 (11.77) | -1.64 (6.53) | -3.47 (8.83)
  Total Score-Youth Variation (n= 56, 57, 23) | -4.71 (9.27) | -4.21 (6.85) | -6.17 (7.71)

11. Secondary Outcome: Change From Baseline in Multidimensional Self Concept Scale (MSCS) at Week 16 Endpoint
Description: The MSCS is an overall assessment of self concept or an individual measure of any of the six scaled dimensions of self concept: Social, Competence, Affect, Academic, Family, and Physical. Standard scores range from 45-145. Higher scores are better (indicate higher self concept).
Time Frame: Baseline, 16 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADHD+ Dyslexia (D): Atomoxetine | ADHD+ Dyslexia (D): Placebo | ADHD Alone: Atomoxetine
Number analyzed (Participants) | 58 | 57 | 25
units on a scale
  Academic Standard Section Score | 5.91 (9.01) | 4.23 (12.77) | 5.52 (6.78)
  Affect Standard Section Score | 3.62 (10.32) | 2.35 (10.81) | 3.56 (10.58)
  Competence Standard Section Score | 6.64 (12.99) | 4.95 (12.05) | 5.20 (9.06)
  Family Standard Section Score | 0.39 (12.52) | -3.12 (11.66) | -1.00 (12.26)
  Physical Standard Section Score | 4.09 (10.34) | 1.32 (12.06) | 3.04 (5.99)
  Social Standard Section Score | 4.36 (11.73) | 2.72 (11.14) | 3.88 (10.39)
  Standard Total Score | 4.72 (9.47) | 1.98 (10.19) | 3.44 (7.70)

12. Secondary Outcome: Change From Baseline in Attention-Deficit/Hyperactivity Disorder Rating Scale (ADHDRS) Total and Subscores - Parent Version at Week 32 Endpoint
Description: The ADHDRS-IV-parent is an 18-item scale with 1 item for each of the 18 symptoms contained in the DSM-IV diagnosis of ADHD. Each item is scored on a 0 to 3 scale: 0=none (never or rarely); 1=mild (sometimes); 2=moderate (often); 3 =severe (very often). Hyperactivity-impulsivity scores range from 0-27, and inattention scores range from 0-27. Total scores range from 0-54. Higher scores indicate higher impairment.
Time Frame: Baseline, 32 weeks
Population: All randomized participants who entered open-label phase with a baseline and at least one post-baseline result, and last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADHD+ Dyslexia (D): Atomoxetine | ADHD Alone: Atomoxetine
Number analyzed (Participants) | 45 | 21
units on a scale
  Hyperactivity-Impulsivity Score | -9.8 (6.17) | -8.29 (4.61)
  Inattention Score | -13.84 (6.56) | -14.33 (7.16)
  Total Score | -23.64 (10.43) | -22.62 (9.07)

13. Secondary Outcome: Change From Baseline in Attention-Deficit/Hyperactivity Disorder Rating Scale (ADHDRS) Total and Subscores - Teacher Version at Week 32 Endpoint
Description: The ADHDRS-IV-Teacher is an 18-item scale with 1 item for each of the 18 symptoms contained in the DSM-IV diagnosis of ADHD. Each item is scored on a 0 to 3 scale: 0=none (never or rarely); 1=mild (sometimes); 2=moderate (often); 3 =severe (very often). Hyperactivity-impulsivity scores range from 0-27, and inattention scores range from 0-27. Total scores range from 0-54. Higher scores indicate higher impairment.
Time Frame: Baseline, 32 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units
Arm/Group | ADHD+ Dyslexia (D): Atomoxetine | ADHD Alone: Atomoxetine
Number analyzed (Participants) | 23 | 9
units
  Hyperactivity-Impulsivity Score | -1.87 (4.80) | -2.89 (4.48)
  Inattention Score | -4.28 (6.08) | -4.19 (4.11)
  Total Score | -6.15 (8.51) | -7.08 (7.34)

14. Secondary Outcome: Change From Baseline in Woodcock-Johnson III Scores at Week 32 Endpoint
Description: as for outcome 4
Time Frame: Baseline, 32 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADHD+ Dyslexia (D): Atomoxetine | ADHD Alone: Atomoxetine
Number analyzed (Participants) | 45 | 21
units on a scale
  Basic Reading Skills (Tests 1, 13 | 2.73 (6.51) | -0.24 (5.37)
  Letter-Word Identification (Test 1) | 1.69 (7.19) | 0.24 (5.73)
  Passage Comprehension (Test 9) | 2.31 (9.18) | 1.24 (5.63)
  Reading Comprehension (Tests 9, 17) | 2.89 (9.07) | 0.86 (7.04)
  Reading Fluency (Test 2) | 2.69 (9.04) | 3.24 (8.64)
  Reading Vocabulary (Test 17) | 2.60 (8.55) | -0.14 (10.57)
  Spelling (Test 7) | 0.60 (7.74) | 0.38 (5.96)
  Spelling of Sounds (Test 20) | 2.98 (10.77) | 5.90 (14.17)
  Word Attack (Test 13) | 3.27 (7.09) | -0.90 (6.59)

15. Secondary Outcome: Change From Baseline in Comprehensive Test of Phonological Processing (CTOPP) at Week 32 Endpoint
Description: as for outcome 5
Time Frame: Baseline, 32 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADHD+ Dyslexia (D): Atomoxetine | ADHD Alone: Atomoxetine
Number analyzed (Participants) | 45 | 21
units on a scale
  Blending Words | 1.31 (2.01) | 1.90 (2.98)
  Elision | 1.07 (2.00) | 0.71 (3.05)
  Memory for Digits | 0.87 (2.17) | -0.05 (2.13)
  Non-word Repetition | 0.93 (2.27) | 0.43 (3.03)
  Phonological Awareness | 7.33 (9.50) | 5.33 (15.99)
  Phonological Memory | 4.93 (10.57) | -0.67 (12.44)
  Rapid Digit Naming | 0.43 (1.91) | 0.62 (2.31)
  Rapid Letter Naming | 0.43 (2.06) | 0.90 (2.34)
  Rapid Naming | 1.30 (11.27) | 1.76 (12.35)

16. Secondary Outcome: Change From Baseline in Gray Oral Reading Test-4 (GORT-4) at Week 32 Endpoint
Description: as for outcome 6
Time Frame: Baseline, 32 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADHD+ Dyslexia (D): Atomoxetine | ADHD Alone: Atomoxetine
Number analyzed (Participants) | 45 | 20
units on a scale
  Accuracy Score | 0.82 (1.30) | 0.95 (1.82)
  Comprehension Score | 0.04 (1.73) | -0.30 (1.59)
  Fluency Score | 0.76 (1.40) | 1.10 (2.63)
  Oral Reading Quotient | 2.64 (15.05) | -1.30 (21.22)
  Rate Score | 0.58 (1.74) | 0.15 (1.98)

17. Secondary Outcome: Change From Baseline in Test of Word Reading Efficiency (TOWRE) at Week 32 Endpoint
Description: as for outcome 7
Time Frame: Baseline, 32 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADHD+ Dyslexia (D): Atomoxetine | ADHD Alone: Atomoxetine
Number analyzed (Participants) | 45 | 21
units on a scale
  Phonemic Decoding Efficiency | 2.64 (6.54) | 5.33 (6.98)
  Sight Word Efficiency | 1.93 (6.51) | 4.62 (8.74)
  Total Word Reading Efficiency Standard Score | 2.56 (17.35) | 1.52 (20.64)

18. Secondary Outcome: Change From Baseline in Working Memory Test Battery for Children (WMTB-C) at Week 32 Endpoint
Description: as for outcome 8
Time Frame: Baseline, 32 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADHD+ Dyslexia (D): Atomoxetine | ADHD Alone: Atomoxetine
Number analyzed (Participants) | 45 | 21
units on a scale
  Phonological Loop Component Score (n=43, 20) | 3.67 (11.27) | 1.70 (9.66)
  Central Executive Component Score (n=38, 14) | 6.53 (11.34) | 1.64 (11.30)
  Visuo-Spatial Sketchpad Component Score (n=40, 20) | 3.85 (12.89) | 2.65 (9.96)
  Digit Recall (n=45, 21) | -0.04 (2.92) | 0.52 (4.08)
  Word List Matching (n=45, 21) | 2.38 (7.96) | 1.95 (8.22)
  Word List Recall (n=45, 21) | 1.49 (3.00) | 0.33 (2.50)
  Non-Word List Recall (n=44, 21) | 0.55 (2.90) | -0.67 (4.39)
  Block Recall (n=45, 21) | 0.71 (3.88) | 1.05 (4.24)
  Mazes Memory (n=45, 21) | 2.33 (7.04) | 3.48 (7.77)
  Listening Recall (n=45, 21) | 2.18 (4.01) | -1.05 (6.42)
  Counting Recall (n=45, 21) | 1.53 (4.65) | 1.24 (6.54)
  Backward Digit Recall (n=45, 21) | 1.07 (3.24) | 2.29 (5.20)

19. Secondary Outcome: Change From Baseline in Life Participation Scale-child (LPS-C) Score at Week 32 Endpoint
Description: as for outcome 9
Time Frame: Baseline, 32 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADHD+ Dyslexia (D): Atomoxetine | ADHD Alone: Atomoxetine
Number analyzed (Participants) | 45 | 21
units on a scale
  LPS Happy/Social Score (n=45, 21) | 1.57 (4.37) | 2.14 (4.30)
  LPS Self Control Score (n=45, 20) | 9.10 (10.73) | 10.44 (10.42)
  LPS Total Score (n=45, 20) | 10.67 (14.27) | 12.64 (13.95)

20. Secondary Outcome: Change From Baseline in Kiddie Sluggish Cognitive Tempo (K-SCT) at Week 32 Endpoint
Description: as for outcome 10
Time Frame: Baseline, 32 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADHD+ Dyslexia (D): Atomoxetine | ADHD Alone: Atomoxetine
Number analyzed (Participants) | 45 | 21
units on a scale
  Total Score-Parent Variation (n=45, 21) | -10.40 (11.94) | -10.83 (10.84)
  Total Score-Teacher Variation (n=23, 9) | -7.00 (12.82) | -7.89 (5.18)
  Total Score-Youth Variation (n=45, 21) | -4.36 (7.57) | -5.43 (8.44)

21. Secondary Outcome: Change From Baseline in Multidimensional Self Concept Scale (MSCS) at Week 32 Endpoint
Description: as for outcome 11
Time Frame: Baseline, 32 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ADHD+ Dyslexia (D): Atomoxetine | ADHD Alone: Atomoxetine
Number analyzed (Participants) | 45 | 21
units on a scale
  Academic Standard Section Score | 6.02 (9.72) | 5.43 (6.98)
  Affect Standard Section Score | 4.29 (11.14) | 3.14 (10.45)
  Competence Standard Section Score | 6.76 (11.77) | 5.19 (7.94)
  Family Standard Section Score | 0.16 (14.40) | 0.33 (9.79)
  Physical Standard Section Score | 6.09 (12.00) | 2.43 (7.20)
  Social Standard Section Score | 4.84 (11.84) | 2.38 (11.75)
  Standard Total Score | 5.61 (10.82) | 3.48 (7.21)

ADVERSE EVENTS:
Arm/Group | Atomoxetine/Atomoxetine | Placebo/Atomoxetine
Serious Adverse Events (participants affected / at risk) | 1/120 | 0/89
Other Adverse Events (participants affected / at risk) | 108/120 | 71/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine/Atomoxetine (N=120) | Placebo/Atomoxetine (N=89)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine/Atomoxetine (N=120) | Placebo/Atomoxetine (N=89)
Abdominal discomfort (Gastrointestinal disorders) | 7 (8) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 23 (31) | 6 (8)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 3 (3)
Nausea (Gastrointestinal disorders) | 34 (42) | 5 (6)
Vomiting (Gastrointestinal disorders) | 16 (24) | 8 (9)
Fatigue (General disorders) | 31 (34) | 9 (11)
Irritability (General disorders) | 14 (15) | 8 (11)
Pyrexia (General disorders) | 2 (3) | 6 (6)
Therapeutic response unexpected (General disorders) | 6 (12) | 2 (2)
Weight decreased (Investigations) | 6 (6) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 22 (22) | 4 (5)
Dizziness (Nervous system disorders) | 15 (16) | 5 (5)
Headache (Nervous system disorders) | 27 (36) | 16 (21)
Somnolence (Nervous system disorders) | 10 (12) | 0 (0)
Aggression (Psychiatric disorders) | 6 (6) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days